CLINICAL TRIAL: NCT00084279
Title: Safety and Tolerability of Consensus Interferon-Alpha (CIFN) Plus Interferon Gamma-1b (IFN-γ 1b) With or Without Ribavirin (RBV) in the Treatment of Patients With Chronic Hepatitis C Who Are Non-Responders to PEG-IFN-a (2a or 2b) Plus RBV
Brief Title: CIFN and IFN γ-1b With or Without Ribavirin for Treatment of Chronic Hepatitis C (Nonresponders)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InterMune (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGHC-002
Record Dates: First submitted 2004-06-09; First posted 2004-06-11 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-07

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Liver; Pegylated; Interferon; Alpha; Gamma; Ribavirin; Combination; Nonresponder; Pegasys; PegIntron
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — interferon gamma-1b; Ribavirin

INTERVENTIONS:
Drug: Consensus Interferon-Alpha, Interferon Gamma-1b, Ribavirin — interferon gamma-1b: 0.25 and 0.5 mL, SQ, 3x per week interferon alfacon: 0.3 mL and 0.5 mL, SQ, once a day Ribavirin: 2 capsules in a.m., 3 capsules in p.m.; daily

SUMMARY:
To evaluate the safety and tolerability of two different doses of Consensus Interferon-Alpha and Interferon Gamma-1b with or without ribavirin in patients with chronic hepatitis C who are non-responders to PEG-IFN-a 2a or PEG-IFN-a 2b plus ribavirin.

ELIGIBILITY:
Inclusion Criteria:

1. Signed, written, informed consent from the patient or legal representative before any study-specific procedures are performed
2. Male or female 18 years of age or older
3. Chronic hepatitis C infection based on history of positive serum anti-HCV antibody and/or HCV RNA
4. Patients must have documented failure to respond to past treatment with PEG-Intron or Pegasys plus RBV.
5. Liver biopsy within 3 years of screening documenting chronic liver disease consistent with chronic hepatitis C

Exclusion Criteria:

1. Patients with any history of decompensated liver disease including but not restricted to portal hypertension as manifested by gastroesophageal varices, variceal bleeding, ascites, or encephalopathy
2. Specific laboratory abnormalities at Screening
3. Patients who were HCV RNA negative during prior pegylated interferon plus ribavirin treatment, but who relapsed during follow-up
4. Recent depression or psychiatric disorders
5. Known HIV infection or positive HIV antibody test at Screening
6. Chronic hepatitis B infection or positive hepatitis B surface antigen (HBsAg) at Screening
7. Unstable or uncontrolled thyroid disease
8. Presence or history of non-HCV chronic liver disease
9. History of unstable or deteriorating cardiovascular or cerebrovascular disease within 6 months prior to Screening
10. Current or history of neurologic disorder within a specified time frame
11. A disease known to cause significant alteration in immunologic function including hematological malignancy, sarcoidosis or autoimmune disorder (e.g. rheumatoid arthritis, systemic lupus erythematosis, leukemia, lymphoma, autoimmune thyroid disease, scleroderma, psoriasis, inflammatory bowel disease, multiple sclerosis etc.)
12. History of major organ transplantation (i.e., liver, kidney, lung, or heart) with an existing functional graft, including bone marrow transplant or stem cell transplant
13. Concurrent therapy with immunosuppressive drugs or cytotoxic agents such as cyclosporine, azathioprine, chronic systemic corticosteroids, or chemotherapeutic agent(s) (e.g., cyclophosphamide, methotrexate, or cancer chemotherapy) or radiation therapy
14. Pregnant or lactating women
15. Liver biopsy within the past three years documenting cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2004-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Virologic response defined as >2 log (base 10) reduction in HCV RNA | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew McClure, MD, Study Director — InterMune
Locations (1):
- InterMune, Inc., Brisbane, California, United States